CLINICAL TRIAL: NCT06616415
Title: A Multicenter, Open-label, Single-arm, Phase 4 Clinical Study to Evaluate the Pharmacokinetics, Efficacy, and Safety of Belumosudil Mesylate Tablets in Chinese Adolescents (Aged From 12 to Less Than 18 Years) With Chronic Graft-versus-host Disease (cGVHD) Who Have Had an Inadequate Response to Glucocorticoids or Other Systemic Therapies
Brief Title: A Clinical Study to Evaluate the Pharmacokinetics, Efficacy, and Safety of Belumosudil in Chinese Adolescents With cGVHD Who Have Had an Inadequate Response to Glucocorticoids or Other Systemic Therapies
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACT18369
Record Dates: First submitted 2024-09-24; First posted 2024-09-27 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Chronic Graft Versus Host Disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — belumosudil; KD025

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Belumosudil (Experimental): Participants will receive belumosudil 200 mg tablets orally QD in 28-day cycles until clinically significant progression of cGVHD
  Interventions: Drug: Belumosudil

INTERVENTIONS:
Drug: Belumosudil — Pharmaceutical form: Tablet Route of administration: Oral
  Other Names: SAR445761/ KD025; Rezurock

SUMMARY:
This is a single group, Phase 4, single-arm post-marketing study for treatment.

The purpose of this study is to verify the pharmacokinetics, efficacy, and safety of belumosudil mesylate tablets in Chinese adolescent participants (aged from 12 to less than 18) with cGVHD who have had an inadequate response to glucocorticoids or other systemic therapies.

Participants will receive treatment with belumosudil tablets 200 mg once daily in 28-day cycles during the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 12 to less than 18 years of age at the time of signing the informed consent.
* Participant has undergone allogeneic hematopoietic stem cell transplantation (allo-HSCT).
* Has active moderate to severe cGVHD.
* Has received at least one line of prior systemic therapy for cGVHD.
* Participant must receive a corticosteroid therapy for cGVHD with a stable dose for at least 2 weeks prior to the first dose of the IMP.
* Has a Lansky-Play performance score of ≥60.
* Participants should have an expected survival of longer than 6 months.
* Body weight of 30 kg and above.
* Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* The participant or their legally authorized representative (LAR) must be capable of giving signed informed consent.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Recurrence of hematologic neoplasms (according to the corresponding criteria for recurrence of primary hematologic neoplasms) or post-transplant lymphoproliferative disease at screening.
* Received investigational systemic therapy for cGVHD within 28 days prior to enrollment, unless the prior treatment had been washed out for at least 28 days or 5 half-lives prior to enrollment, whichever is shorter.
* Absolute neutrophil count (ANC) <1.0 × 10^9/L.
* Platelet count <50 × 10^9/L.
* Alanine aminotransferase (ALT) >3× the upper limit of normal (ULN), aspartate aminotransferase (AST) >3 × ULN.
* Total bilirubin (TBIL) >1.5 × ULN (>3 ULN if Gilbert's syndrome).
* Estimated Glomerular Filtration Rate (eGFR) <30 mL/min/1.73 m^2 using the revised Bedside Schwartz formula . Revised Schwartz equation: CrCl (mL/min/1.73 m^2) = 0.413 × (height [in cm])/Creatinine (in mg/dL) at screening visit.
* Participant not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions, or participants potentially at risk of noncompliance to study procedures.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2024-12-04 (Actual); Primary Completion 2026-05-13 (Estimated); Study Completion 2026-05-13 (Estimated)

PRIMARY OUTCOMES:
Plasma concentrations of belumosudil at specified time points | At Day 1 and Day 29(±3)

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 18 month
  Overall response rate (ORR, including complete response [CR] and partial response [PR]), which will be assessed by the investigator according to the NIH Consensus Criteria (2014) at any time before the start of new systemic treatment for cGVHD.
Duration of response (DoR) | Up to 18 month
  Duration of response (DoR): time from the date of the first response to the date of cGVHD progression as defined by 2014 NIH consensus response criteria, start of new systemic treatment for cGVHD, or death, whichever occurs first. DOR is determined only for participants who achieved overall response (PR or CR) as per 2014 NIH consensus response criteria.
System organ response rate | Up to 18 month
  System organ response rate: proportion of participants who achieve an overall response (CR or PR) for each of the nine individual organs (Skin, Eyes, Mouth, Esophagus, Upper GI, Lower GI, Liver, Lungs, and Joints and fascia) as per 2014 NIH consensus response criteria at any time before the start of new systemic treatment for cGVHD
Number and proportion of participants with dose reduction in corticosteroid during the treatment period | Up to 18 month
Failure-free survival (FFS) | Up to 18 month
  Failure-free survival (FFS): time from the date of the first administration of IMP to 1) the date of initiation of new systemic treatment for cGVHD, or 2) date of death, or 3) date of recurrent underlying disease, whichever occurs first
Overall survival (OS) | Up to 18 month
  Overall survival (OS): time from the date of the first administration of IMP to the date of death due to any cause
Change in cGVHD severity based on physician-reported overall cGVHD activity | Up to 18 month
Change in symptom activity assessed based on patient-reported cGVHD activity | Up to 18 month
Modified Lee cGVHD Symptom Scale change | Up to 18 month
  The scale contains 30 items grouped in 7 subscales (skin, eye, mouth, lung, nutrition, energy, and psychological). Patients report how "bothered" they feel about each symptom using a five-point Likert scale from "not at all" (0) to "extremely" (4). A higher score indicating worse symptoms, reporting score will be normalizing to a 0 to 100 scale.
Number and proportion of participants with calcineurin inhibitor (CNI) dose reduction or discontinuation during the treatment period | Up to 18 month
Number of participants with treatment-emergent adverse events (TEAEs), serious TEAEs, and adverse events of special interest (AESIs) | Up to 18 month

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- China (2):
  - Investigational Site Number : 1560001, Beijing
  - Investigational Site Number : 1560002, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org